CLINICAL TRIAL: NCT04372498
Title: An Explananatory, Proof-of-concept Study of Senicapoc in Patients With Familial Dehydrated Stomatocytosis Caused by the V282M Mutation in the Gardos (KCNN4) Channel
Brief Title: Senicapoc and Dehydrated Stomatocytosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Carlo Brugnara, Director of the Hematology Laboratory, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-P00034327
Record Dates: First submitted 2020-04-30; First posted 2020-05-04 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Dehydrated Hereditary Stomatocytosis
MeSH Terms: conditions — Xerocytosis, hereditary | interventions — senicapoc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): This is a pivotal trial in members of the same family carrying the V282M nutation in the Gardos channel (KCNN4) and other patients with V282 mutations with demonstrated in-vitro sensitivity to senicapoc. These mutations lead to hyperactivation of the channel and red cell dehydration. Up to 6 patients are eligible to enroll in this study, which will assess effectiveness based on individual changes of primary endpoints over individually established baselines.
  Interventions: Drug: Senicapoc (synonyms: ICA-17043; 2,2-bis-(4-fluorophenyl)-2-phenylacetamide)

INTERVENTIONS:
Drug: Senicapoc (synonyms: ICA-17043; 2,2-bis-(4-fluorophenyl)-2-phenylacetamide) — This study is conducted as open label, with each patient's response determined with an adaptive Bayesian model based on historical and baseline values for the primary endpoints of the trial. 3 monthly dose escalation steps will assess the efficacy of senicapoc in a dose range (10-40 mg/day) which has been used in prior trials for other indications.

SUMMARY:
Dehydrated stomatocytosis is a genetic disorder characterized by chronic hemolysis, variable anemia and erythrocyte dehydration. Causative mutations have been identified in either the Gardos (KCNN4) channel or the mechanosensitive channel PIEZO1. Senicapoc is a selective blocker of the Gardos channel that has been extensively studied in sickle cell disease and shown to be safe with limited side-effects. However, senicapoc did not meet the designated clinical endpoints in a pivotal phase 3 trial. The present study is an explanatory, proof-of-concept study of Senicapoc administered once daily in patients with familial dehydrated stomatocytosis caused by autosomal dominant V282 mutations in the Gardos (KCNN4) channel.

DETAILED DESCRIPTION:
The proposed study is an explanatory, proof-of-concept study of Senicapoc administered once daily in patients with familial dehydrated stomatocytosis caused by the autosomal dominant V282 mutation in the Gardos (KCNN4) channel. The study population will include up to 6 members of the same family, all carrying the V282M mutation, and other V282 mutations with demonstrated in-vitro sensitivity to senicapoc, meeting study criteria for inclusion and exclusion. Patients will begin the study with a loading dose of 20 mg/day for 4 days followed by a dose of 10 mg once daily for the first 4 weeks of study.

After 4 weeks at the initial dose, patients will be escalated to higher doses (in 3 steps of 10 mg every 4 weeks) to a maximal dose of 40 mg once daily.

Patients who demonstrate response in the primary endpoints at the end of the efficacy study, and who have not been permanently discontinued due to Senicapoc-attributed serious adverse events (SAE), will be eligible for a 12-month study extension at the dose determined to be effective in the treatment efficacy study.

Patients who meet inclusion criteria will be enrolled at visit 0, and if available, will be provided with the appropriated instrument to record daily pain scores and other QOL indicators. Treatment will begin at Visit 1, which will follow visit 0 after 2-3 weeks. After an effective dose and tolerated has been established in the dose escalation period, patients will be seen every two weeks until they reach 24 weeks of treatment. Patients will be seen for a potential maximum of 19 visits in the treatment efficacy phase of the study, with additional phone contacts after the first week of treatment and within a week from each dose escalation.

At the end of the efficacy portion of the study, patients will be eligible to participate in a one-year optional open-label extension, provided that they have not been permanently discontinued from the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients carrying KCNN4 mutations in V282M as described in 1981 by Snyder et al and Sauberman et al. and characterized molecularly by Andolfo et al. in 2015 , and other patients with V282 mutations with demonstrated in-vitro sensitivity to senicapoc, will be eligible to participate in this study if they meet all the following criteria:

  1. Have a diagnosis of dehydrated stomatocytosis with a molecularly confirmed mutation in KCNN4.
  2. Are at least 21 years of age.
  3. Have hematological manifestations of dehydrated stomatocytosis such as elevated MCHC, compensated or uncompensated chronic hemolysis, with reticulocytosis. For enrollment, 3/5 of the following baseline value must meet enrollment criteria:

     Reference Range Enrollment criterion MCHC 32-36 mg/dL > 36 mg/dL Reticulocyte count (absolute) 0.25-0.90 x 103/µL > 0.200 x 103/µL Bilirubin, Indirect 0.2-1.2 mg/dL > 1.5 mg/dL Haptoglobin. 43-212 mg/dL < normal LDH 100-220 U/L > normal
  4. Personally dated and signed informed consent detailing all the pertinent aspects of the study.
  5. Willingness to adhere to study visit schedule, treatment plan, blood draws and laboratory tests and other study procedures.

Exclusion Criteria:

* Patient will be excluded from the study if they meet any of the following criteria:
* RBC transfusion in the prior 90 days.
* Recent (within the past 30 days) hospitalization for major surgical procedure, infection requiring IV treatment, or significant bleeding complications.
* Recent (within 2 weeks) diagnosis of cerebrovascular accident of transient ischemic attack.
* Hepatic dysfunction serum alanine transferase or GGT values > 3 times the upper limit of normal, total serum bilirubin values > 20 mg/dL
* Renal disease (defined as serum creatinine greater than 1.2 mg/dL, or a requirement for chronic dialysis).
* Severe symptomatic anemia defined as a Hct value < 18%.
* Any other severe acute or chronic medical condition or laboratory alteration that may increase the risks associated with participation to this study and/or administration of senicapoc, based on the clinical judgement of the principal investigator.
* Any condition that may interfere with the study subject's ability to adhere to study schedule, or comply with blood drawing requirements, such as inadequate venous access.
* Pregnancy or breastfeeding for female subjects.
* Concurrent use of illicit drugs and/or alcohol dependence, as determined by the principal investigator.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
chronic hemolysis biomarkers | 6 months
  Reticulocyte count, bilirubin, LDH, Hemoglobin

SECONDARY OUTCOMES:
Decrease in the frequency and intensity of pain | 6 months
  Splenic, abdominal or other, assessed with Numeric Pain Rating Scale (NPRS).
Improved functional health and well-being | 6 months
  FACT-An QOL questionnaire
Decrease in the frequency and intensity of pain | optional, 6 months
  patient diaries or PDA
spleen volume | if available, 6-months
  three-dimensional ultrasonography

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Brugnara, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andolfo I, Russo R, Manna F, Shmukler BE, Gambale A, Vitiello G, De Rosa G, Brugnara C, Alper SL, Snyder LM, Iolascon A. Novel Gardos channel mutations linked to dehydrated hereditary stomatocytosis (xerocytosis). Am J Hematol. 2015 Oct;90(10):921-6. doi: 10.1002/ajh.24117. PMID 26178367
- [Background] Snyder LM, Sauberman N, Condara H, Dolan J, Jacobs J, Szymanski I, Fortier NL. Red cell membrane response to hydrogen peroxide-sensitivity in hereditary xerocytosis and in other abnormal red cells. Br J Haematol. 1981 Jul;48(3):435-44. doi: 10.1111/j.1365-2141.1981.tb02735.x. PMID 7259992
- [Background] Sauberman N, Fairbanks G, Lutz HU, Fortier NL, Snyder LM. Altered red blood cell surface area in hereditary xerocytosis. Clin Chim Acta. 1981 Aug 10;114(2-3):149-61. doi: 10.1016/0009-8981(81)90388-0. PMID 7285342